CLINICAL TRIAL: NCT02704923
Title: Atropine for Preventing Ventilator-Associated Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Responsible Party: Principal Investigator, Cassiano Mateus Forcelini, Professor, PhD, MD, Universidade de Passo Fundo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAAE 40374815.3.0000.5342
Record Dates: First submitted 2016-02-26; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Ventilator-Associated Pneumonia
Keywords: Atropine; Pneumonia; Ventilator; Adults; Intensive care unit.
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Pneumonia | interventions — Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atropine (Active Comparator)
  Interventions: Drug: Atropine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atropine — Atropine eye drops (1%) administered by sublingual way (2 drops) every 6 hours
  Other Names: Atropine eye drops
  Arms: Atropine
Drug: Placebo — Placebo eye drops characterized by saline administered by sublingual way (2 drops) every 6 hours
  Other Names: Placebo eye drops
  Arms: Placebo

SUMMARY:
A double-blind, placebo controlled trial of atropine eye drops used by sublingual way for preventing Ventilator-Associated Pneumonia.

DETAILED DESCRIPTION:
A double-blind, placebo controlled trial of atropine eye drops used by sublingual way for preventing Ventilator-Associated Pneumonia was conducted in Passo Fundo - RS, south Brazil. 40 adult patients were included (exploratory stage 2 trial). Interventions were initiated until 48 hours of patients were submitted to orotracheal intubation: 2 drops of atropine (eye drop) by sublingual way, compared to placebo on the same regimen. Efficacy outcomes were pneumonia and death, but safety was also assessed. No difference was observed between the placebo and atropine groups in terms of efficacy and safety outcomes. The small sample and a significance difference in terms of initiating the interventions (medians: 48h for atropine; 24h for placebo) may be a conservative bias. This can not exclude a possible benefit of atropine that should be better evaluated in a stage 3 trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted in intensive care unit with endotracheal intubation and ventilator initiated until 48 hours

Exclusion Criteria:

* Pneumonia, radiotherapy, chemiotherapy, conditions that interfere with saliva production or change normal oral cavity shape

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Ventilator-Associated Pneumonia | through the end of the study, an average of one year
  Incidence of ventilator-associated pneumonia through the end of the study, an average of one year

SECONDARY OUTCOMES:
Death | through the end of the study, an average of one year
  Incidence of death through the end of the study, an average of one year

OTHER OUTCOMES:
Adverse events | through the end of the study, an average of one year
  Incidence of adverse events through the end of the study, an average of one year

IPD SHARING:
Plan to Share IPD: No